CLINICAL TRIAL: NCT07143968
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial of Resmetirom for the Treatment of Metabolic Dysfunction- Associated Steatotic Liver Disease (MASLD) in People Living With Human Immunodeficiency Virus (HIV)
Brief Title: A Study to Evaluate the Use of Resmetirom in Participants With MASLD and HIV
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Naga P. Chalasani (Other)
Responsible Party: Sponsor-Investigator, Naga P. Chalasani, Professor of Medicine, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HCRN005
Record Dates: First submitted 2025-08-25; First posted 2025-08-27 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; HIV (Human Immunodeficiency Virus)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — resmetirom

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Resmetirom - 80mg or 100mg based on participant weight
  Interventions: Drug: Resmetirom
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Drug: Resmetirom — Resmetirom - 80mg or 100mg based on participant weight
  Arms: Treatment
Drug: Placebo Control — Placebo - an identical looking tablet with no medicinal properties
  Arms: Placebo

SUMMARY:
The purpose of this research study is to test the safety and effectiveness of the study drug, resmetirom, in participants with MASLD and HIV. This is a research study to test a drug that is already on the market with a population that was not included in the original clinical trials. Participants will be people over age 18 with HIV who are on antiretroviral therapy and have been diagnosed with MASLD.

Researchers will compare resmetirom to placebo (a look-alike substance that contains no drug) to see if resmetirom decreases the amount of fat in the liver.

Participants will:

* Complete 3 screening visits to determine eligibility.
* Take resmetirom or placebo every day for 24 weeks if eligible.
* Have 2 MRI scans to measure the amount of fat on the liver. One will be before treatment starts and one will be at the end of 24 weeks of treatment.
* Attend 3 scheduled clinic visits while on treatment for bloodwork and safety assessments.
* Participate in 3 phone calls while on treatment and one phone call 4 weeks after treatment is completed to check for safety and any health changes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years of age) with documented HIV.
2. Documented diagnosis of MASLD established by imaging (ultrasound, CT scan or MRI) or vibration-controlled transient elastography (VCTE) or liver biopsy within 12 months before screening.
3. Hepatic fat fraction ≥8% by MRI-PDFF.
4. Liver stiffness by VCTE ≥8 kPa and CAP≥263 dB/m
5. HIV-1 RNA <200 copies/mL for ≥6 months on antiretroviral therapy (ART) (must have screening HIV-1 RNA value and one clinical care value within 6 months prior to screening and up to the randomization that meet the criteria).
6. Stable ART regimen for ≥3 months prior to screening and stable up to the randomization and no active plans to change ART while on study.
7. Willingness to participate in the study.

Exclusion Criteria:

1. History of significant alcohol consumption (defined as >2 drinks/day on average for men, >1 drinks/day on average for women) for at least 3 consecutive months (12 consecutive weeks) within 5 year before screening
2. History of other acute or chronic liver disease, including, but not limited to autoimmune, primary biliary cholangitis, Wilson's disease, alpha 1 antitrypsin deficiency, hemochromatosis, hepatitis B virus (HBV), and ongoing or recent (within the past 3 years) hepatitis C RNA positivity.
3. History of liver transplant.
4. Liver biopsy or radiologic imaging consistent with the clinical presence of cirrhosis or portal hypertension at screening.
5. Participants whose Visit 2 ALT, AST, or alkaline phosphatase (ALP) values exceed their Visit 1 values by more than 50%.
6. Inability to undergo MRI testing
7. Uncontrolled T2DM defined as glycated hemoglobin (HbA1c) >9.5% at screening.
8. Any of the following laboratory values at screening:

   1. ALT or AST >250 U/L.
   2. Total bilirubin (TBL) >1.5 mg/dL and direct bilirubin > 0.5 mg/dL (unless due to Gilbert's disease or atazanavir use, per the opinion of the site investigator).
   3. Platelet count <150,000/mm3.
   4. Estimated glomerular filtration rate (e-GFR) <60 mL/min/1.73m2 using the chronic kidney disease-epidemiology collaboration (CKD-EPI) equation
   5. International normalized ratio (INR) >1.3.
   6. Albumin < 3.6 g/dL
9. Liver stiffness measurement (LSM) by VCTE > 20 kPa
10. Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in hepatic fat content at week 24 | From baseline to the end of treatment at 24 weeks

SECONDARY OUTCOMES:
Proportion of participants with reduction of at least 30% in hepatic fat content from baseline to week 24 | Baseline to the end of treatment at week 24
Change from baseline in liver enzyme parameters, lipid profile and fasting glucose | From baseline to end of treatment at week 24

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Alabama Birmingham, Birmingham, Alabama
  - UC San Diego Altman Clinical and Translational Research Institute, La Jolla, California
  - University of California, San Francisco, San Francisco, California
  - Atlantic Clinical Research Institute, West Palm Beach, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Mt Sinai Health System, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - UT Health Houston, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided
Await IRB determination of privacy and HIPAA issues